CLINICAL TRIAL: NCT05046847
Title: Phase I Clinical Study to Evaluate the Tolerability and Pharmacokinetics of TQB3811 Tablets in Patients With Advanced Malignant Tumors
Brief Title: A Clinical Study to Evaluate the Tolerability and Pharmacokinetics of TQB3811 Tablets in Patients With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3811-I-01
Record Dates: First submitted 2021-09-13; First posted 2021-09-16 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3811 (Experimental): The initial dose is 2.5mg, once a day (QD), and the medication stage is divided into single administration and continuous administration. The single administration is given once a day, and the continuous administration is entered 4 days after drug withdrawal. The drug is administered continuously until the disease progresses.
  Interventions: Drug: TQB3811

INTERVENTIONS:
Drug: TQB3811 — TQB3811 is a second-generation TrkA inhibitor.

SUMMARY:
TQB3811 tablet is a second-generation tropomyosin receptor kinase (TRK) inhibitor that selectively inhibits the kinase activity of TRKA, TRKB, and TRKC, and also selectively inhibits the kinase activity of TRKA, TRKB, and TRKC that produce secondary drug-resistant mutations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced malignancy diagnosed histologically and/or cytologically, who have failed standard treatment or are unable to receive standard treatment or have no effective treatment.
* Age: 18~75 years old.
* Women of childbearing age must be negative for serum or urine HCG within 7 days prior to study enrollment and must be non-lactating; Patients should agree to use contraception during the study period and for 6 months after the study period.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months.
* Patients voluntarily joined the study and signed the informed consent, showing good compliance.

Exclusion Criteria:

* Patients has had or is currently having other malignant tumors within 3 years.
* Patients have multiple factors that affect their oral medication (such as inability to swallow, chronic diarrhea, and intestinal obstruction).
* The patient had unmitigated toxic reactions due to any prior treatment.
* Patients underwent major surgical treatment, open biopsy, or significant traumatic injury within 4 weeks prior to the start of study treatment.
* Patients have long-term unhealed wounds or fractures.
* The patient had experienced an arterial/venous thrombosis event in the past 6 months, such as a cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis, and pulmonary embolism.
* The patient has a history of psychotropic drug abuse and cannot quit or has mental disorders.
* Patients are taking cytochrome P450 3A (CYP3A) inhibitors or inducers.
* Patients have uncontrolled pleural effusion, pericardial effusion, or ascites that still require repeated drainage.
* Patients with brain metastases with symptoms or control of symptoms for less than 2 weeks.
* The patients were currently breastfeeding or planned to breastfeed during the study period.
* Patients who, in the investigator's judgment, have a comorbidity that seriously endangers patient safety or interferes with study completion, or who are considered unsuitable for inclusion for other reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline up to 32 weeks
  To evaluate MTD of TQB3811 tablets in Chinese adult patients with advanced solid tumors
Adverse events (AEs) and serious adverse events (SAEs) | Baseline up to 28 days
  The occurrence of all AEs and SAEs
Dose-limiting toxicity (DLT) | Baseline up to 32 weeks
  To evaluate DLT of TQB3811 tablets in Chinese adult patients with advanced solid tumors

SECONDARY OUTCOMES:
Time to reach maximum (peak) plasma concentration following drug administration（Tmax） | 15, 30minutes, 1, 2, 4, 6, 8,10, 24, 48 hours after oral administration of day 1 and day 11;30 minutes before oral administration on day 1, day5, day7,day8 ,day 9 and day11.
  To characterize the pharmacokinetics of TQB3811 by assessment of time to reach maximum plasma concentration after single and multiple dosing
Maximum (peak) plasma drug concentration （Cmax） | 15, 30 minutes, 1, 2, 4, 6, 8,10, 24, 48 hours after oral administration of day 1 ;30 minutes before oral administration on day 1.
  Cmax is the maximum plasma concentration of TQB3811 or metabolite(s).
Elimination half-life （t1/2） | 15, 30minutes, 1, 2, 4, 6, 8,10, 24, 48 hours after oral administration of day 1 and day 11;30 minutes before oral administration on day 1, day5, day7,day8 ,day 9 and day11.
  t1/2 is time it takes for the blood concentration of TQB3811 or metabolite(s) to drop by half.
Area under the plasma concentration-time curve from time zero to time t （AUC0-t） | 15, 30 minutes, 1, 2, 4, 6, 8,10, 24, 48 hours after oral administration of day 1 ;30 minutes before oral administration on day 1.
  To characterize the pharmacokinetics of TQB3811 by assessment of area under the plasma concentration time curve from the first dose to infinity.
Maximum (peak) steady-state plasma drug concentration during a dosage interval （Cmax,ss） | 15, 30 minutes, 1, 2, 4, 6, 8,10, 24, 48 hours after oral administration of day 1 and day 11;30 minutes before oral administration on day 1, day5, day7,day8 ,day 9 and day11.
  Cmax,ss is maximum (peak) steady-state plasma drug concentration during a dosage interval .
Minimum steady-state plasma drug concentration during a dosage interval （Css-min） | 15, 30 minutes, 1, 2, 4, 6, 8,10, 24, 48 hours after oral administration of day 1 and day 11;30 minutes before oral administration on day 1, day5, day7,day8 ,day 9 and day11.
  Css-min is minimum steady-state plasma drug concentration during a dosage interval.
Concentration at the end of the dosing interval (AUCtau,ss) | 15, 30 minutes, 1, 2, 4, 6, 8,10, 24, 48 hours after oral administration of day 1 and day 11;30 minutes before oral administration on day 1, day5, day7,day8 ,day 9 and day11.
  To characterize the pharmacokinetics of TQB3811 by assessment of area The concentration at the end of the administration interval
Progress Free Survival（PFS） | up to 96 weeks
  From the start of randomization to the first tumor progression or time of death.
Disease control rate（DCR） | up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Response (DOR) | up to 96 weeks
  The time when the participants first achieved complete or partial remission to disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China